CLINICAL TRIAL: NCT06986603
Title: Glucagon Dose-Response in Patients With Post-Bariatric Hypoglycemia
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Virginia (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00000270; R01DK137518 (NIH)
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hypoglycemia; Hypoglycemia, Reactive; Bariatric Surgery
Keywords: glucagon sensitivity
MeSH Terms: conditions — Hypoglycemia | interventions — Glucagon; Injections

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either increasing doses of glucagon or decreasing doses of glucagon for visit 3, and the other during visit 4.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ascending doses of glucagon (Experimental): Participants will receive sequential ascending doses of glucagon, 75, 150, 300, 450 micrograms during the course of the study visit.
  Interventions: Drug: Glucagon for Injection (Fresenius Kabi USA)
- descending doses of glucagon (Experimental): Participants will receive sequential descending doses of glucagon - 300, 150, 75 micrograms
  Interventions: Drug: Glucagon for Injection (Fresenius Kabi USA)

INTERVENTIONS:
Drug: Glucagon for Injection (Fresenius Kabi USA) — We are assessing response to glucose, including incremental glucose values as well as changes in endogenous glucose production, insulin secretion, and glucagon levels.

SUMMARY:
The purpose of the study is to determine how blood sugar levels in individuals with and without hypoglycemia after bariatric surgery respond to different doses of glucagon, a hormone that is usually present in your body that regulates blood sugar levels. In this study, there will be 4 visits to the clinical research center. In the first visit, medical history and physical exam will be performed, and blood samples will be taken to assess overall health. During visit 2, a continuous glucose monitor will be placed under the skin. (This may be combined with visit 1, depending on the schedule of visits.) In visit 3, we will test the effect of a total of 4 different doses of glucagon, in increasing doses. In visit 4, we will test the effect of a total of 3 doses of glucagon, in decreasing doses. For both visit 3 and 4, we will infuse labeled stable glucose to allow us to measure how much glucose the body is making, and will measure levels of hormones which regulate glucose, such as insulin and glucagon.

DETAILED DESCRIPTION:
Visit 1 (Screening) This visit will last about 2 hours.

You will be instructed to come to Joslin Diabetes Center after fasting for at least 8 hours (nothing but water for eight hours before your visit).

During the screening visit, a study team member will go over the informed consent form with you and they will help explain why this study is being done and the study procedures involved. You will have to sign the consent form before any study related procedures take place. After you sign the consent, the following tests and procedures will be done to ensure you are eligible and it is safe for you to continue study participation. These include the following:

* Review medical history and medications. There are certain medications that you may not be able to take during the study. Any changes to your medications will be reviewed with the study doctor and information will be provided to you in writing.
* Physical examination and vital signs (blood pressure, heart rate, temperature, height and weight).
* Blood tests (about one tablespoon of blood) to check your blood counts, liver and kidney tests and blood sugar
* Urine test to check for pregnancy (if you are a female of child bearing potential) that must be negative in order to continue participation.
* Surveys regarding frequency and symptoms of your low blood sugar levels (hypoglycemia)
* If you experience low blood sugars (hypoglycemia), we will ask you to complete a log including information about: prior meal, exercise (if any), what symptoms you experienced, how you treated it, and blood sugar at that moment if you checked it.
* An Electrocardiogram (ECG or EKG) will be performed.
* You will have some sticky patches applied to your chest and sometimes your arms and legs to help record electrical activity of you heart.
* Each sticky patch has a wire that is attached to a monitor.
* The ECG will only take a few minutes to complete; you need to lie still on your back until the ECG is completed.

Any changes to your medications will be reviewed with the study doctor and will be provided to you in writing.

The study team will give you a phone call once the results of this visit are available to notify you whether you are eligible or not for the study. If these tests show you are eligible, you will be scheduled to report to Joslin Diabetes Center for the CGM visit.

Visit 2 (CGM Placement) This visit will last up to 1 hour and will occur within 7-10 days before Visit 3. This visit may be combined with your screening visit, depending on scheduling needs.

If you are already using a CGM, you will skip this visit and you will continue using your CGM as you were previously doing. If you were not previously using a CGM, you will come to Joslin Diabetes Center. You will receive a continuous glucose monitor (CGM) that will allow us to track your glucose throughout the day and night, including highs and lows. This device is approved by the FDA, and it will be paid for by the study. A small sensor will be placed just underneath the skin of your abdomen or on the back of your upper arm with the help of a plastic needle so that glucose can be measured every 5 minutes. However, CGM will be used in "masked" mode for the entire duration of the study, which means that you will not be able to see sugar levels or receive alerts if you have high or low blood sugars. This is just used to record your blood sugar during the study. You will need to check your blood sugar by the finger stick method frequently while the CGM is in place. You should check your fingerstick whenever you have symptoms of low blood sugar. If you have episodes of low blood sugar (hypoglycemia), you will be asked to complete a log of the food and drinks you consumed. You will also add to the log: time and severity of any symptoms of low blood sugar, exercise (if any), and fingerstick glucose levels if you check them. The CGM only lasts 10 days, so if all visits are not completed in this time frame, the CGM will need to be replaced. At the end of the study (all study visits) the CGM will be removed.

Randomization:

The glucagon dosing pattern during the study will be randomly decided - as by the flip of a coin. You will be randomized into starting with the increasing dose arm or the decreasing dose arm. You may decide if you wish to return to complete the second dose arm or not. For example, if you are randomized into the increasing dose arm, after completion of the study visit, you may return if you wish to complete the decreasing dose study arm. You may wish to participate in one or both study visits 3 and 4. Your participation in visit 4 is completely optional.

Visit 3 (Glucagon) This visit will last approximately 5 hours.

A study team member will call you one day prior to the study day to inform you that if you experience low blood sugar in the night before your admission, we will need to reschedule your study visit to another day. You will arrive at Joslin Diabetes Center at around 7AM after fasting overnight for at least 8 hours (i.e., no food/calories after 11 PM the night before). The study team will record your blood pressure, heart rate, temperature, weight, medications you are taking and collect a urine sample from you for a pregnancy test (if applicable).

You will have one IV catheter placed in the vein of your forearm (near the elbow).

Another IV will be started in the back of your hand or forearm in the other arm. This IV will be used for drawing blood periodically during the study.

An IV catheter is a thin tube inserted into the vein using a needle. Once the catheter is in place, the needle is removed but the tube remains in the vein. The needle is replaced by a small cap above the tube, which allows blood to be drawn from the vein and for agents to be administered through it.

The IV in your forearm will have a "stable" or cold glucose (sugar) tracer (meaning that there is no radiation involved) infused in very small amounts throughout the duration of the study visit. These are naturally occurring substances present in your body and they behave exactly the same as regular sugar. The glucose tracer is necessary to measure and track how much glucose is made in your body during the study duration. There is no known risk of stable tracers of glucose.

The IV in the back of your hand, will rest in a see-through box ('hotbox') that is heated and will make drawing blood samples from this vein easier, and your blood sugar levels and hormones will be measured every five to ten minutes from this IV.

Starting at approximately 10 am, small doses of glucagon (hormone naturally present in your body to control your blood sugar levels) will be injected just under the skin of your belly or arm every half hour either from low to medium dose or medium to low dose, depending on the randomization above, for a total of three or four doses. The dose of glucagon will be increased or decreased gradually but the total dose injected (975 or 525 micrograms) during the entire study visit will not exceed the maximum allowable dose (1000 micrograms) for treatment of low blood sugar.

* An infusion of nonradioactive stable glucose tracer will be started through the vein at approximately 8 AM and continued until the end of the study.
* An IV (plastic tube) will be inserted into one of your hands for blood draw.
* The hand will then be placed in a heated plexiglass box (at about 55 C°) to enable periodic blood draws during this time.
* Small doses of glucagon will be injected under the skin every half hour for a total of four doses
* Following the last blood draw, all infusions will be stopped and all IV catheters will be removed.

During this study visit, you will not be allowed to get out of bed or use the commode for about four hours because such activities could disconnect the infusion catheters and disturb data collection. You will be offered use of bedpan/bottle or, only if necessary, an in and out urinary catheter. A urinary catheter is a thin, flexible tube that is inserted into the bladder and collects urine into a drainage bag.

If you decide to participate in visit 4, and the CGM will not last until that visit, we will replace the CGM as described above, before you are discharged from the Clinical Research Unit. If you are not participating in visit 4, this will be your last visit of the study and the CGM will be removed at the end of this visit.

Visit 4 (Glucagon) This visit will last approximately 5 hours and will take place within 7-10 days of visit 3.

This visit will be identical to visit 3, except that the dose of glucagon will be reversed from medium to low and only three doses of glucagon will be injected every half hour. The order of the visits will be decided randomly like the flip of a coin as described above.

To summarize,

• If you complete the entire study, you will be in the study for up to 6 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-70 years of age, inclusive, at screening.
2. Willingness to provide informed consent and follow all study procedures, including attending all scheduled visits.
3. Males or females diagnosed with ongoing PBH, at least 2 years following Roux-en-Y gastric bypass (RYGB), with documented episodes of hypoglycemia, and history of fulfillment of Whipple's triad.

Exclusion criteria:

1. Documented hypoglycemia occurring only in the fasting state (>12 hours fast);
2. Current diabetes, defined as hemoglobin A1c >6.5% or use of diabetes medications, except for acarbose or miglitol;
3. Chronic kidney disease stage 4 or 5 (including end-stage renal disease);
4. Hepatic disease, including serum ALT or AST greater than 2 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0;
5. Congestive heart failure, NYHA class II, III or IV;
6. History of myocardial infarction, unstable angina or revascularization within the past 6 months.
7. Two or more risk factors for coronary artery disease including diabetes, uncontrolled hypertension, uncontrolled hyperlipidemia, and active tobacco use.
8. History of recurrent syncope (unrelated to hypoglycemia) or active diagnosis of a cardiac arrhythmia;
9. Current administration of β-blocker therapy;
10. History of a cerebrovascular accident;
11. Seizure disorder (other than with suspect or documented hypoglycemia);
12. Active treatment with long-acting (LAR) octreotide or pasireotide;
13. Active malignancy, except basal cell or squamous cell skin cancers;
14. Personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma (MEN 2, neurofibromatosis, or Von Hippel-Lindau disease);
15. Known insulinoma;
16. Major surgical operation within 30 days prior to screening;
17. Clinically significant anemia as defined as a hematocrit < 33%;
18. Bleeding disorder, treatment with warfarin, or platelet count <50,000;
19. Blood donation (1 pint of whole blood) within the past 2 months;
20. Active alcohol abuse or substance abuse;
21. Current administration of oral or parenteral corticosteroids;
22. Pregnancy and/ or lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test before any procedures.
23. Not enrolled in another study that uses an investigational drug for this condition.

    -

    Exclusion Criteria:

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Incremental change in plasma glucose levels after administration of exogenous glucagon for each dose. | Measurement of glucose levels will occur at baseline, and then every 5 minutes, for 60 minutes.
  Glycemic response to exogenous glucagon for doses, as measured by incremental change in plasma glucose levels at each 30 minute step of the dose escalation protocol. AUC will be compared in each of the 2 study visits (escalation vs. deescalation).
Endogenous glucose production (EGP) after administration of exogenous glucagon. | Measurement of glucose levels will occur at visit 2, at baseline, and then every 5 minutes after the first dose of glucagon, for 120 minutes
  Response to exogenous glucagon as measured by the incremental change in EGP from baseline during dose escalation or deescalation protocol.

SECONDARY OUTCOMES:
Incremental change in plasma insulin levels during glucagon dose escalation protocol | Measurement of insulin levels will occur at baseline, and then every 30 minutes after each dosetes.
  Insulin response to exogenous glucagon, as measured by incremental change in plasma insulin during dose escalation protocol
Insulin secretion rate in response to exogenous glucagon | Measurement of insulin secretion rates will occur at visit 2, at baseline, and then 30 minutes after each dose of glucagon
  Insulin secretion rate in response to exogenous glucagon, as measured using the C-peptide model
Incremental change in GLP1 levels during glucagon dosing protocol | Measurement will occur at visit 2, at baseline, and then every 30 minutes after each dose of glucagon
  GLP1 response to exogenous glucagon, as measured by incremental change in GLP1

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - Joslin Diabetes Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Only deidentified information will be shared.